CLINICAL TRIAL: NCT05207358
Title: Minimizing Glucocorticoid Administration in Patients With Proliferative Lupus Nephritis During the Induction of Remission Period-EUROLUPUS vs. RITUXILUP Regimen: A Randomized Study
Brief Title: Minimizing Glucocorticoid Administration in Patients With Proliferative Lupus Nephritis
Acronym: GLUREDLUP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Institutul Clinic Fundeni (Other)
Responsible Party: Principal Investigator, Bogdan Obrisca, Assist. Prof., Institutul Clinic Fundeni
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FundeniCI
Record Dates: First submitted 2021-12-07; First posted 2022-01-26 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Lupus Nephritis
Keywords: immunosuppression; glucocorticoids; eurolupus; rituxilup; induction therapy
MeSH Terms: conditions — Lupus Nephritis | interventions — Rituximab; Mycophenolic Acid; Cyclophosphamide; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RITUXILUP regimen (Experimental): - 2 doses of Rituximab 1 g and Methylprednisolone 500 mg on days 1 and 15. Patients will receive Mycophenolate Mofetil, initially 500 mg twice daily, titrated to a maximum of 1.5 g twice daily, depending on leukocyte count and digestive tolerance, which will be maintained 24 months.
  Interventions: Drug: Rituximab; Drug: Mycophenolate Mofetil
- EUROLUPUS regimen (Standard therapy) (Other): 3 daily pulses of 750 mg of intravenous Methylprednisolone, followed by oral corticosteroid therapy starting with a dose of 0.5 mg / kg / day for 4 weeks, then decreased by 2.5 mg of Prednisolone / day each 2 weeks. A low dose of glucocorticoid (5-7.5 mg / day) is maintained until 24 months after enrollment. All patients will receive Cyclophosphamide intravenously starting day 1, 6 pulses at a fixed dose of 500 mg given at 2 weeks. After 3 months, Azathioprine (2 mg / kg / day) is initiated 2 weeks after the last administration of Cyclophosphamide and maintained for the next 21 months.
  Interventions: Drug: Cyclophosphamide; Drug: Corticosteroids

INTERVENTIONS:
Drug: Rituximab — 2 doses of Rituximab 1 g and Methylprednisolone 500 mg on days 1 and 15.
  Arms: RITUXILUP regimen
Drug: Mycophenolate Mofetil — Patients will receive Mycophenolate Mofetil, initially 500 mg twice daily, titrated to a maximum of 1.5 g twice daily, depending on leukocyte count and digestive tolerance, which will be maintained 24 months.
  Arms: RITUXILUP regimen
Drug: Cyclophosphamide — All patients will receive Cyclophosphamide intravenously starting day 1, 6 pulses at a fixed dose of 500 mg given at 2 weeks. After 3 months, Azathioprine (2 mg / kg / day) is initiated 2 weeks after the last administration of Cyclophosphamide and maintained for the next 21 months.
  Arms: EUROLUPUS regimen (Standard therapy)
Drug: Corticosteroids — 3 daily pulses of 750 mg of intravenous Methylprednisolone, followed by oral corticosteroid therapy starting with a dose of 0.5 mg / kg / day for 4 weeks, then decreased by 2.5 mg of Prednisolone / day each 2 weeks. A low dose of glucocorticoid (5-7.5 mg / day) is maintained until 24 months after enrollment.
  Arms: EUROLUPUS regimen (Standard therapy)

SUMMARY:
The aim of the study is to evaluate the efficacy of a therapeutic regimen which decreases glucocorticoid exposure compared with standard therapy in patients with proliferative lupus nephritis during remission induction by evaluating the histological and clinical remission.

DETAILED DESCRIPTION:
After an initial screening phase during which a first kidney biopsy is performed, all patients that meet the inclusion criteria will be randomized to one of the treatment arms:

* EUROLUPUS regimen: 3 daily pulses of 750 mg of intravenous Methylprednisolone, followed by oral corticosteroid therapy starting with a dose of 0.5 mg / kg / day for 4 weeks, then decreased by 2.5 mg of Prednisolone / day each 2 weeks. A low dose of glucocorticoid (5-7.5 mg / day) is maintained until 24 months after enrollment. All patients will receive Cyclophosphamide intravenously starting day 1, 6 pulses at a fixed dose of 500 mg given at 2 weeks. After 3 months, Azathioprine (2 mg / kg / day) is initiated 2 weeks after the last administration of Cyclophosphamide and maintained for the next 21 months.
* RITUXILUP regimen: 2 doses of Rituximab 1 g and Methylprednisolone 500 mg on days 1 and 15. Patients will receive Mycophenolate Mofetil, initially 500 mg twice daily, titrated to a maximum of 1.5 g twice daily, depending on leukocyte count and digestive tolerance, which will be maintained 24 months.

Second kidney biopsy will be performed 6 months after the start of the treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Age of the patient between 18 and 80 years,
* Patients diagnosed with systemic lupus erythematosus according to ACR 1997 or SLICC-2012 criteria
* Diagnosis of proliferative lupus nephritis class III, IV +/- V (confirmed by renal biopsy and classified according to ISN / RPS);
* Estimated glomerular filtration rate by CKD-EPI> 30 ml / min / 1.73 sqm
* Estimated glomerular filtration rate by CKD-EPI <30 ml / min / 1.73 sqm but> 15 ml / min / 1.73 sqm with chronicity index (according to NIH score) <6
* Absence of contraindications to the use of Methylprednisolone, Mycophenolate mofetil, oral corticosteroids or Rituximab
* Ability to provide informed consent

Exclusion Criteria:

* The patient's age under 18 years
* Patients with life-threatening complications (e.g. Cerebritis)
* Estimated glomerular filtration rate by CKD-EPI <30 ml / min / 1.73 sqm
* Estimated glomerular filtration rate by CKD-EPI <30 ml / min / 1.73 sqm but> 15 ml / min / 1.73 sqm with chronicity index (according to NIH score)> 6
* Presence of pregnancy / lactation
* Patients who have received more than 2 g of Methylprednisolone intravenously in the last 4 weeks
* Use in the last 3 months of biological therapy
* Use of intravenous immunoglobulins / plasmapheresis in the last 6 months
* The presence of an active infection
* History of neoplasia
* Comorbidities requiring systemic corticosteroid therapy
* Non-adhesion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with a histological remission | 6 months
  The primary endpoint is to evaluate the histologic remission at 6 months after initiation of induction treatment assessed by the change in the individual active lesions and in the activity modified NIH score.

SECONDARY OUTCOMES:
Percentage of participants with a complete renal response | 12 months
  Complete renal response is defined by the combination of a decrease in proteinuria below 500 mg / g Creatinine, an inactive urinary sediment and a return of serum Creatinine to baseline.
Percentage of patients with severe infectious episodes effects | 24 months
Cumulative exposure to glucocorticoids | 24 months
The proportion of patients who obtained a complete renal response | 6, 18 and 24 months
The proportion of patients who obtained a partial renal response | 6, 12, 18, 24 months
  Partial renal response is defined as a 50% decrease in proteinuria (if the proteinuria was nephrotic the decrease is defined as a 50% reduction in proteinuria to values <3000 mg / g) and stabilization (+/- 25%) or decrease, but not normalization of serum Creatinine.
The proportion of patients who have developed relapse | 24 months
Proportion of patients who showed normalization of complement fractions C3, C4 and negative anti-dcDNA antibodies at week 52 | 52 weeks
Proportion of patients with progression of chronicity score by more than 2 units | 6 months
  Evaluation of the histologic progression at 6 months after initiation of induction treatment assessed by the change in the individual chronic lesions and in the chronicity modified NIH score.
Percentage of patients with non-severe infectious episodes | 24 months
Percentage of patients with severe non-infectious adverse events | 24 months
Percentage of patients with non-severe non-infectious adverse events | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Gener Ismail, MD, PhD, Principal Investigator — Institutul Clinic Fundeni
Locations (1):
- Fundeni Clinical Institute, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 12 months of publishing the results of the primary endpoints of the study

REFERENCES:
- [Background] Parikh SV, Almaani S, Brodsky S, Rovin BH. Update on Lupus Nephritis: Core Curriculum 2020. Am J Kidney Dis. 2020 Aug;76(2):265-281. doi: 10.1053/j.ajkd.2019.10.017. Epub 2020 Mar 24. PMID 32220510
- [Background] Pepper R, Griffith M, Kirwan C, Levy J, Taube D, Pusey C, Lightstone L, Cairns T. Rituximab is an effective treatment for lupus nephritis and allows a reduction in maintenance steroids. Nephrol Dial Transplant. 2009 Dec;24(12):3717-23. doi: 10.1093/ndt/gfp336. Epub 2009 Jul 17. PMID 19617257
- [Background] Fanouriakis A, Bertsias G. Changing paradigms in the treatment of systemic lupus erythematosus. Lupus Sci Med. 2019 Feb 8;6(1):e000310. doi: 10.1136/lupus-2018-000310. eCollection 2019. PMID 31168398
- [Background] Parikh SV, Rovin BH. Current and Emerging Therapies for Lupus Nephritis. J Am Soc Nephrol. 2016 Oct;27(10):2929-2939. doi: 10.1681/ASN.2016040415. Epub 2016 Jun 9. PMID 27283496
- [Background] Catapano F, Chaudhry AN, Jones RB, Smith KG, Jayne DW. Long-term efficacy and safety of rituximab in refractory and relapsing systemic lupus erythematosus. Nephrol Dial Transplant. 2010 Nov;25(11):3586-92. doi: 10.1093/ndt/gfq256. Epub 2010 May 11. PMID 20466686
- [Background] Rovin BH, Furie R, Latinis K, Looney RJ, Fervenza FC, Sanchez-Guerrero J, Maciuca R, Zhang D, Garg JP, Brunetta P, Appel G; LUNAR Investigator Group. Efficacy and safety of rituximab in patients with active proliferative lupus nephritis: the Lupus Nephritis Assessment with Rituximab study. Arthritis Rheum. 2012 Apr;64(4):1215-26. doi: 10.1002/art.34359. Epub 2012 Jan 9. PMID 22231479
- [Background] Tamirou F, Houssiau FA. Management of Lupus Nephritis. J Clin Med. 2021 Feb 9;10(4):670. doi: 10.3390/jcm10040670. PMID 33572385
- [Background] Condon MB, Ashby D, Pepper RJ, Cook HT, Levy JB, Griffith M, Cairns TD, Lightstone L. Prospective observational single-centre cohort study to evaluate the effectiveness of treating lupus nephritis with rituximab and mycophenolate mofetil but no oral steroids. Ann Rheum Dis. 2013 Aug;72(8):1280-6. doi: 10.1136/annrheumdis-2012-202844. Epub 2013 Jun 5. PMID 23740227
- [Background] Morales E, Galindo M, Trujillo H, Praga M. Update on Lupus Nephritis: Looking for a New Vision. Nephron. 2021;145(1):1-13. doi: 10.1159/000511268. Epub 2020 Nov 4. PMID 33147587
- [Background] Bajema IM, Wilhelmus S, Alpers CE, Bruijn JA, Colvin RB, Cook HT, D'Agati VD, Ferrario F, Haas M, Jennette JC, Joh K, Nast CC, Noel LH, Rijnink EC, Roberts ISD, Seshan SV, Sethi S, Fogo AB. Revision of the International Society of Nephrology/Renal Pathology Society classification for lupus nephritis: clarification of definitions, and modified National Institutes of Health activity and chronicity indices. Kidney Int. 2018 Apr;93(4):789-796. doi: 10.1016/j.kint.2017.11.023. Epub 2018 Feb 16. PMID 29459092